CLINICAL TRIAL: NCT01058447
Title: An Open, Single-Dose, Single-Centre, Phase I Study to Assess the Metabolism, Excretion and Pharmacokinetics of [14C]AZD1981 in Healthy Male Volunteers
Brief Title: Study to Assess the Metabolism, Excretion and Pharmacokinetics of [14C]AZD1981 in Healthy Male Volunteers
Acronym: ADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D9830C00006
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: ADME; Healthy volunteers
MeSH Terms: interventions — AZD1981

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD1981

INTERVENTIONS:
Drug: AZD1981 — Oral tablet, 250 mg, single dose

SUMMARY:
The purpose of the study is to characterize the absorption, distribution, metabolism and excretion (ADME) of a single oral dose of [14C]AZD1981

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedure
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Exposed to radiation levels above background of >5 mSv in the last year, >10 mSv over the last 5 years or a cumulative total of >1 mSv per year of life
* History or presence of any clinically significant disease or disorder in the opinion of the investigator
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline in the opinion of the investigator

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables and Radioactivity | Frequent sampling occasions during study days

SECONDARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab) | Frequent sampling occasions during study days

CONTACTS AND LOCATIONS:
Overall Officials: Eva S Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Tim Mant, Professor, Principal Investigator — Quintiles Drug Research Unit at Guy´s Hospital, London, United Kingdom